CLINICAL TRIAL: NCT03565757
Title: Feasibility and Acceptability of a Stress Management and Resilience Training (SMART) Intervention for Family Caregivers of Individuals With Advanced Cancer Undergoing Outpatient Chemotherapy
Brief Title: Stress Management and Resilience Training (SMART) Intervention for Family Caregivers of Individuals With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sherry S. Chesak, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-006696
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Family Caregivers; Advanced Cancer
Keywords: Stress Management; Resilience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART intervention (Experimental): 90-minute SMART small group session
  Interventions: Behavioral: SMART intervention

INTERVENTIONS:
Behavioral: SMART intervention — All participants will attend a 90-minute SMART small group session. This session provides education on the stress response and the principles of gratitude, compassion, mindful presence, and resilient mindset. In addition to the class, there will be follow-up online and written resources.

SUMMARY:
This study examines Stress Management and Resilience Training (SMART) for family caregivers (FCG) of patients receiving chemotherapy for advanced cancer to potentially help with the stressful aspects of providing care. All participants will receive the SMART intervention.

DETAILED DESCRIPTION:
FCGs experience stress and extensive demands in providing care for those with head and neck cancer. Teaching the principles of mindfulness and compassion to FCGs has the potential to protect their psychological health and well-being. This may allow them to provide effective, compassionate care to patients, which ultimately puts the needs of the patient first.

Mindfulness interventions have demonstrated decreased stress and anxiety, and improved self-compassion for individuals, but entail numerous sessions over several weeks, a barrier for caregivers. The SMART program, a brief mindfulness program, has demonstrated improvements in resilience, anxiety, perceived stress, and mindfulness for healthcare providers and patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of patient with advanced head and neck cancer receiving chemotherapy, living with the patient at least 50% of the time during treatment, able to read and speak English, cognitively intact, able to take SMART class within 2 weeks of enrollment

Exclusion Criteria:

* Self-identified mental health diagnoses, less than 18 years of age, not living with patient at least 50% of the time, unable to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Satisfaction score at 8 weeks | Week 8
  The Was It Worth It (WiWi) questionnaire measures satisfaction in seven questions. The questions are answered as either "yes, no, or unsure," overall perception of life change and experience, an open-ended response question, and an option to talk with someone about concerns. Positive responses will indicate acceptability; results reported as individual items.
Change in Mean Self Compassion Scale-Short Form Score at 8 weeks | Baseline and Week 8
  The Self Compassion Scale-Short Form will measure self-compassion. This form includes 12 items that are measured on a 4-point scale from "never" to "very often" with higher score indicating a higher level of perceived stress; some of these items are scored in reverse.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Chesak, PhD, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials